CLINICAL TRIAL: NCT06505083
Title: The Effect of Modified Stepping Trainings in Frailty Elderly With Physical Performance- a Prospective Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonticha Kaewjoho (Other)
Collaborators: Mae Fah Luang University (Other); University of Phayao (Other)
Responsible Party: Sponsor-Investigator, Chonticha Kaewjoho, Department of Allied Health Sciences, University of Phayao
Organization: University of Phayao (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UPhayaoChonticha-218
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-07

CONDITIONS: Rehabilitation; Training; Respiratory Muscle Strength
Keywords: balance ability; gait training; risk of falls; community-dwelling; older adults

STUDY DESIGN:
Intervention Model Description: This prospective randomized controlled trial design was conducted in thirty-two community-dwelling older participants who completed a modified stepping exercises program for 50 minutes/day, three days/week over six weeks. They were assessed for their functional mobility relating to levels of independence and prospectively followed up periods one month.
  RESULTS: The participants in our study demonstrated significant improvements in their functional mobility after within 4 weeks of training, and these improvements continued to increase by week 6 (p<0.01). Notably, the participants showed significant improvements in all functional outcomes at week 4, week 6, and one-month follow-up (p<0.05). The most significant improvements were observed in the FTSST, TUGT, and lower limb muscle strength, and these outcomes were significantly different from the pre-test and intermediate tests (p<0.01).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control grops (Sham Comparator): stepping on stable step
  Interventions: Other: modified stepping trainings
- experimental group (Experimental): stepping on unstable step
  Interventions: Other: modified stepping trainings

INTERVENTIONS:
Other: modified stepping trainings — step-up on box texture difference
  Other Names: stable stepping; unstable stepping

SUMMARY:
This single-blind, randomized controlled trial compared the effects of modifiled stepping exercise training on flat step and unstable step on the functional outcomes in community-dwelling older adults. The subjects were involved in a step up in 4 directions exercise on each surface, according to their groups, for 50 min/day, 3 days/week, for 6 weeks. The functional outcomes were assessed prior to training, at Week 3, Week 6 after training and 1 months after training.

ELIGIBILITY:
Inclusion Criteria:

* The eligible participants needed ability of independent walking over at least 10 m without any assistive devices, and did not participate in a regular exercise program prior to being involved in the study. Older individuals who presented any signs and symptoms that might affect walking and the ability to participate in the study, such as unstable medical conditions, inflammation in the joints of the lower extremities (with a pain scale of more than 5 out of 10 on a visual analog scale), and having sequelae of neurological deficits, were excluded from the study

Exclusion Criteria:

* people who were initially recruited, those diagnosed with dementia, depression, severe cardiovascular disease, or mental illness were excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Timed up and go test (TUGT) | pre test, 4 week, 6 week, 1 month follow up
  The study subjects were instructed to sit on a chair (46cm height) without arm rest. They were instructed to get up from chair on command, walk at a comfortable pace, walk around the cone which was marked 3m ahead and return to a seated position on the original chair. The stop watch was started as soon as the subject lifted buttocks off the chair and it was stopped at the point where the subject sat back in the chair after completing walking. The total time taken by each subject to complete the task was noted as the final score
The five-times-sit-to-stand (FTSTS) test | pre test, 4 week, 6 week, 1 month follow up
  a simple and quick test initially designed to be a proxy measure of lower-limb strength. The test requires a subject to stand up and sit down five times as quickly as possible from a chair with a seat 43-cm high. The time taken to complete the test (the FTSTS scores) is recorded with a stopwatch. Excellent test-retest reliability of FTSTS scores (intraclass correlation coefficient (ICC) 0.933) has been reported in people with chronic stroke and community-dwelling older adults (ICC 0.89- 0.96). Several other studies have demonstrated the reliability or validity or both of FTSTS scores in specific subject populations, including Parkinson's disease (Duncan et al., 2011) and renal pathologies and subjects with rheumatoid arthritis and balance disorders

SECONDARY OUTCOMES:
Individual isometric muscle strength | pre test, 4 week, 6 week, 1 month follow up
  The strength of maximum isometric voluntary contraction of the subject's hip flexor, extensor, adductor, abductor, knee flexor, extensors, ankle dorsiflexors, and plantar flexors (in kilograms) was measured using a Nicholas handheld dynamometer (model 01,160, Lafayette Instrument Company, Lafayette, IN). The Nicholas HHD is a digital force gauge capable of measuring forces from 0.0 to 199.99 kg. The measurement protocol was as described by (Magalhães et al., 2012)
Back-leg-chest strength | pre test, 4 week, 6 week, 1 month follow up
  A calibrated BLC dynamometer (The Takei 5402 Back Muscle Digital Dynamometer) measures isometric muscle strength, recorded in kilograms (kg) of force. There is excellent test-retest reliability (ICC = .98) for leg extension strength (Ten Hoor et al., 2016). The dial ranges from 0 to 300 kg (0 to 660 lb) in 10 kg (10 lb) increments. For the test, the length of the chain was adjusted to the participants' height by asking the subject to stand on the base of the BLC dynamometer with extended knees. Subsequently, the handle was positioned at the height of the intra-articular space of the knee joint. For the test, participants had to stand on the base, with knees and hips flexed slightly while the lower back had to maintain an appropriate lordotic curve.
The 10-m Walk Test (10-m WT) | pre test, 4 week, 6 week, 1 month follow up
  This test generally evaluates the gait velocity of patients with neurological damage and shows high inter-rater and intra-rater reliability (r=0.89-1.00) (Lang et al., 2016; Saito et al., 2022). In the present study, the subjects were instructed to individuals performed three 10-m overground walk trials timed with a stopwatch in each comfortable and maximum speeds to characterize our participant sample. For comfortable walking speed, individuals were instructed to "walk at a speed that feels the most comfortable" and for maximum speed individuals were instructed to "walk at the fastest speed you feel safe" walk 10 m; the time taken for 4 m, excluding the first 3 m and the last 3 m, which take into account acceleration and deceleration, was measured in units of seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Mar Fah Luang university, Chiang Rai, Chiangrai, Thailand